CLINICAL TRIAL: NCT00245908
Title: ASTHMA (AntibioticS To Help Manage Asthma) Pilot Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wisconsin Research Network (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC Protocol 98-370-277
Record Dates: First submitted 2005-10-27; First posted 2005-10-28 (Estimated); Last update posted 2005-10-28 (Estimated); Status verified 2002-01

CONDITIONS: Asthma
Keywords: Asthma; Chlamydia pneumoniae; Chlamydophila pneumoniae; Azithromycin
MeSH Terms: conditions — Asthma | interventions — Azithromycin

INTERVENTIONS:
Drug: azithromycin

SUMMARY:
The ASTHMA Pilot Study is a randomized, controlled, parallel group clinical trial of 6 weekly doses of azithromycin (cumulative dose 4800 mg) or placebo as adjunctive treatment in addition to usual care for adults with stable persistent asthma, with final follow up at 3 months after completion of study medication.

The hypothesis to be tested is that antibiotic treatment will improve asthma at followup, and that this improvement will be limited to patients with evidence of C. pneumoniae infection.

The secondary hypothesis is that randomized, controlled treatment trials can be carried out successfully in a geographically dispersed practice-based research network.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory bronchial condition of unknown etiology. Decades ago many clinicians believed that infection played a major role in asthma etiology, but current expert opinion favors the view that asthma is a noninfectious condition whose root cause is inflammation. Therefore chronic antiinflammatory therapy, mainly inhaled corticosteroids, is currently advocated as primary anti-asthma treatment. It is important to recognize, however, that antiinflammatory therapy is palliative, not curative.

A growing body of evidence implicates chronic bronchial infection with Chlamydia pneumoniae in the pathogenesis of asthma in both adults and children. Organism identification studies (culture and PCR) suggest that up to one-half of children with asthma may be chronically infected by C. pneumoniae, and seroepidemiologic studies in adults are consistent with chronic C. pneumoniae infection in the majority of adult-onset asthmatics. Furthermore, case reports and uncontrolled trials have provided provocative but inconclusive evidence that treatment of C. pneumoniae infection in both children and adults with asthma can favorably affect the natural history of this disorder.

We propose a randomized, placebo-controlled, triple-blinded study of antichlamydial antimicrobial therapy in adult-onset asthma. Results will help to determine whether antimicrobial therapy is effective in treating some adult asthma syndromes. Positive results would have significant public health implications. Methodologies developed for use in this trial may expedite future studies in practice-based research networks.

ELIGIBILITY:
Inclusion Criteria:

* adults with stable persistent asthma and evidence for reversible airway obstruction

Exclusion Criteria:

* macrolide allergy, pregnancy or lactation, specified comorbidities or medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 1999-09; Study Completion 2002-09

PRIMARY OUTCOMES:
None specified (pilot study)
Clinical outcomes measured: asthma symptoms, medication use, asthma-specific qulaity-of-life
Serological measures: Chlamydia pneumonaie IgG, IgA by ELISA at baseline and follow up

CONTACTS AND LOCATIONS:
Overall Officials: David L Hahn, MD, MS, Principal Investigator — Wisconsin Research Network

REFERENCES:
- [Background] Hahn DL, Plane MB. Feasibility of a practical clinical trial for asthma conducted in primary care. J Am Board Fam Pract. 2004 May-Jun;17(3):190-5. doi: 10.3122/jabfm.17.3.190. PMID 15226283